CLINICAL TRIAL: NCT06873620
Title: Impact of the Cardiopulmonary Bypass and Cross-Clamp Time Ratio on Postoperative Outcomes in Open Heart Surgery: A Prospective Observational Analysis
Status: Completed | Type: Observational
Sponsor: Ahmet Yuksek (Other Government)
Responsible Party: Sponsor-Investigator, Ahmet Yuksek, Associate Professor, Kocaeli City Hospital
Organization: Kocaeli City Hospital (Other Government)
Other Study IDs: KSH-2024-23
Record Dates: First submitted 2025-03-07; First posted 2025-03-12 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: CABG; Cardiac Anesthesia; Cardiac Surgery Prognosis; Bypass Complication; On-pump Valve Surgery or CABG; Anesthesia
Keywords: on-pump cabg; cardiac anesthesia; cross clamping; cabg complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- on-pomp CABG: All eligible patients undergoing on-pump-assisted CABG surgery will be included in this group.

SUMMARY:
This study aims to investigate the relationship between the ratio of cardiopulmonary bypass (CPB) time to cross-clamp (CC) time and postoperative complications in open heart surgery. While CPB time and CC duration have been linked to complications, no study has explored the specific ratio between CPB time and CC time in relation to postoperative outcomes. This prospective study seeks to fill that gap.

DETAILED DESCRIPTION:
Open heart surgery involves several distinct stages: 1) preparation for cardiopulmonary bypass (CPB), 2) the CPB phase, which includes the cross-clamp (CC) process, and 3) hemostasis and closure. During the CPB phase, the left internal mammary artery (LIMA) and saphenous vein are freed for coronary anastomosis, followed by arterial and venous cannulation. Once cannulation is completed, CPB is initiated. A cross-clamp is placed on the aorta to stop the heart, and cardioplegia solution is administered. Afterward, distal anastomoses are performed, and once completed, the cross-clamp is removed and the heart begins to beat again. The duration the cross-clamp remains in place is referred to as the CC time. In the CPB phase, proximal anastomoses are made on the aorta. After checking for any bleeding, thoracic drains are placed, and the CPB is terminated. Once all controls are in place, the chest is closed, and the patient is transferred to the intensive care unit.

The mortality rate for open heart surgery varies between 1% and 5%, depending on the patient's specific characteristics. Postoperative complications such as bleeding revision, acute kidney injury, liver failure, respiratory failure, and heart failure are common. Literature has linked these complications to vascular conditions, CPB time, and the duration of cross-clamp time. However, no studies were found that specifically compare the ratio of CPB time to CC time with postoperative complications.

In this study, we aim to prospectively investigate the relationship between the ratio of CPB time to cross-clamp time and postoperative complications in patients undergoing open heart surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing open heart surgery
* Undergo on pump surgery

Exclusion Criteria:

* Patients undergoing emergency open heart surgery Patients undergoing open heart surgery on a beating heart

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will be an observational research conducted in our hospital, involving patients aged 18 to 80 who are undergoing on-pump coronary artery bypass grafting (CABG). The study population will consist of individuals within this age range who are scheduled for elective or urgent on-pump CABG surgery.
Sampling Method: Non-Probability Sample
Enrollment: 348 (Actual)
Dates: Start 2024-02-23 (Actual); Primary Completion 2025-10-01 (Actual); Study Completion 2025-10-15 (Actual)

PRIMARY OUTCOMES:
Relationship between CPB/CC time and mortality | From enrollment to the end of treatment at 8 weeks
  CPB/CC time is the ratio of cardiopulmonary bypass (CPB) time to cross-clamp (CC) time in patients undergoing on-pump cardiac surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet Yilmaz, Associate Proffessor, Principal Investigator — Kocaeli City Hospital
Locations (1):
- Kocaeli City Hospital, Kocaeli, Izmit, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Sharing IPD is at the discretion of the institution and written permission must be applied to the institution.

REFERENCES:
- [Background] Yousefshahi F, Samadi E, Paknejad O, Movafegh A, Barkhordari K, Bastan Hagh E, Dehestani B. Prevalence and Risk Factors of Hypoxemia after Coronary Artery Bypass Grafting: The Time to Change Our Conceptions. J Tehran Heart Cent. 2019 Apr;14(2):74-80. PMID 31723349
- [Background] Moh'd AF, Al-Odwan HT, Altarabsheh S, Makahleh ZM, Khasawneh MA. Predictors of aortic clamp time duration and intensive care unit length of stay in elective adult cardiac surgery. Egypt Heart J. 2021 Oct 22;73(1):92. doi: 10.1186/s43044-021-00195-0. PMID 34677684
- [Background] Parmana IMA, Boom CE, Rachmadi L, Hanafy DA, Widyastuti Y, Mansyur M, Siswanto BB. Correlation Between Cardiac Index, Plasma Troponin I, Myocardial Histopathology, CPB and AoX Duration in Glutamine versus No Glutamine Administered Patients with Low Ejection Fraction Undergoing Elective On-Pump CABG Surgery: Secondary Analysis of an RCT. Vasc Health Risk Manag. 2023 Feb 28;19:93-101. doi: 10.2147/VHRM.S399925. eCollection 2023. PMID 36880009
- [Background] Hadipourzadeh F, Rastravan R, Totonchi Z, Heydarpur E, Faritous Z. Evaluating the relationship between lactate levels during coronary artery bypass graft surgery and postoperative renal dysfunction. J Cardiovasc Thorac Res. 2024;16(2):129-134. doi: 10.34172/jcvtr.33051. Epub 2024 Jun 25. PMID 39253341